CLINICAL TRIAL: NCT02582385
Title: In-situ Cytokines Expression in the CNS in Amyotrophic Lateral Sclerosis
Brief Title: In-situ Cytokines Expression in the CNS in Amyotrophic Lateral Sclerosis (ALS)
Status: Completed | Type: Observational
Sponsor: Brugmann University Hospital (Other)
Responsible Party: Principal Investigator, Carine DE PREZ, Head of clinic, Brugmann University Hospital
Other Study IDs: CHUB-ALS
Record Dates: First submitted 2015-10-20; First posted 2015-10-21 (Estimated); Last update posted 2015-10-21 (Estimated); Status verified 2015-10

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: Amyotrophic lateral sclerosis (ALS); Cytokines; Neuropathology
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Archived/residual histopathology sections and paraffin blocks entirely from residual autopsy material. Archived material involves old cases (autopsied between 2000 and 2005). All autopsies were conducted within the legal frame of the then applicable laws. There is no reference whatsoever to names or identifications of the deceased patients (anonymous samples).
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Amyotrophic lateral sclerosis (ALS): Archived/residual histopathology sections and paraffin blocks, retrieved entirely from residual autopsy material from patients who died with an amyotrophic lateral sclerosis.
  Interventions: Other: in-situ cytokine expression
- Control: Archived/residual histopathology sections and paraffin blocks, retrieved entirely from residual autopsy material from one non-ALS case.
  Interventions: Other: in-situ cytokine expression

INTERVENTIONS:
Other: in-situ cytokine expression

SUMMARY:
The investigators aim at exploring the differential/topographical in-situ expression of cytokines in the central nervous system (CNS) of patients who died with amyotrophic lateral sclerosis (ALS), using archived histopathology slides and residual paraffin blocks from autopsied cases. Previous studies from the investigators and other groups showed that inflammatory cytokines are implicated in several neurological affections, particularly neurodegenerative conditions. However, in-situ cytokine expression has never been studied so far in ALS. The investigators wanted to see if these neuro-mediators are involved in the neuromolecular chain/cascade underlying ALS.

ELIGIBILITY:
Inclusion Criteria:

* patients who died with amyotrophic lateral sclerosis, having been autopsied.

Exclusion Criteria:

* N/A

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Archived/residual histopathology slides and paraffin blocks from residual autopsy material from patients who died with amyotrophic lateral sclerosis.
Sampling Method: Non-Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2012-10; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
in situ cytokine detection: interleukin 18 | retrospective study performed on archived paraffin blocks, autopsies performed between 2000 and 2005
  IHC detection on histopathology sections of paraffin embedded brain tissue.
in situ cytokine detection: interleukin 1 | retrospective study performed on archived paraffin blocks, autopsies performed between 2000 and 2005
  IHC detection on histopathology sections of paraffin embedded brain tissue.
in situ cytokine detection: interleukin 6 | retrospective study performed on archived paraffin blocks, autopsies performed between 2000 and 2005
  IHC detection on histopathology sections of paraffin embedded brain tissue.
in situ cytokine detection:TNF-a | retrospective study performed on archived paraffin blocks, autopsies performed between 2000 and 2005
  IHC detection on histopathology sections of paraffin embedded brain tissue.

CONTACTS AND LOCATIONS:
Overall Officials: Hazim Kadhim, MD, PhD, Principal Investigator — CHU Brugmann
Locations (1):
- CHU Brugmann, Brussels, Belgium